CLINICAL TRIAL: NCT04648605
Title: Post-traumatic Stress Disorder Occurrence in Parents of Neonate and Children Hospitalized in an Intensive Care Unit
Brief Title: Post-traumatic Stress Disorder After Pediatric Intensive Care Unit Hospitalization
Acronym: POETIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/20/0406
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Post-traumatic Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Questionary (Experimental): Questionary for all parents
  Interventions: Other: Post traumatic stress disorder questionnaire

INTERVENTIONS:
Other: Post traumatic stress disorder questionnaire — Parents of hospitalized children in pediatric resuscitation carry out a validated questionnaire that validates the post-traumatic stress level by a score.

SUMMARY:
The elements that promote the development of post-traumatic stress in parents following hospitalization in pediatric resuscitation and thus the options for improving initial care at the time of hospitalization are unknown.

It is therefore important to describe the prevalence of post-traumatic stress disorder with current pediatric resuscitation management data, but also to possibly describe the factors associated with it in order to optimize initial management.

ELIGIBILITY:
Inclusion Criteria:

- All parents of children aged 0 to 18 who have been admitted in paediatric resuscitation unit.

Exclusion Criteria:

* Holders of parental authority who cannot answer the questionnaire because they do not speak French.
* Opposition of one of the two holders of parental authority
* Minor parental authority holders
* Holders of parental authority under safeguarding of justice or guardianship

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 87 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of post-traumatic stress disorder among parents of newborns, infants and children who have been hospitalized in a paediatric resuscitation unit. | Between one and 6 months after hospitalization.
  Parents will complete Post-traumatic stress disorder Checklist. We will consider subjects with a score above 44 to be clinically affected by post-traumatic stress disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie BREINIG, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France